CLINICAL TRIAL: NCT00672594
Title: Investigator-Initiated Pilot Study of Sunitinib Malate in Patients With Newly Diagnosed Prostate Cancer Prior to Prostatectomy
Brief Title: Study of Sunitinib Malate in Patients With Newly Diagnosed Prostate Cancer Prior to Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007396; DUMC-8725 (Other: Duke legacy protocol number)
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-05

CONDITIONS: Prostate Cancer; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib Malate (Experimental): Sunitinib Malate 50mg capsule by mouth once daily for 4 weeks
  Interventions: Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Sunitinib Malate — Sunitinib Malate 50mg capsule by mouth once daily for 4 weeks
  Other Names: Sutent

SUMMARY:
The purpose of this study is to look at blood and tissue samples for changes following the use of Sunitinib malate. Additionally, we would like to find out if the drug, Sunitinib malate, is safe and works in men with prostate cancer. Sunitinib malate , also known as Sutent, is approved by the U.S. Food and Drug Administration (FDA), for treatment of tumors of intestines and kidney but it is being tested in research studies for use in men with prostate cancer.

DETAILED DESCRIPTION:
Eligible patients will be treated with 50 mg once daily for four weeks followed by one to two weeks off treatment prior to undergoing radical prostatectomy. Patients with palpable disease (cT2-3) and patients with 3 or more positive prostatic biopsies from one lobe may undergo an additional study of IFP monitoring before treatment and during week 4 of study treatment. Safety and tolerability of Sunitinib malate therapy at this dose and schedule in this patient population will be assessed. Extensive correlative science evaluations, including assessment of physiologic, cellular, molecular and genetic changes during treatment with Sunitinib malate, will be performed

ELIGIBILITY:
Inclusion Criteria:

* Histologic evidence of adenocarcinoma of the prostate deemed candidates for curative RRP
* Intermediate or high risk, clinically localized disease
* Adequate organ function
* Patients must be surgically sterile or must agree to use effective contraception during the period of therapy
* Select imaging to rule out metastasis will be done as clinically indicated
* Signed and date informed consent document

Exclusion Criteria:

* Prior treatment for prostate cancer
* Major surgery or radiation therapy within 4 weeks of starting the study treatment
* NCI CTCAE grade 3 hemorrhage within 4 weeks of starting therapy
* History of or known metastatic prostate cancer
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE grade 2 or greater
* QTc interval > 500 msec on baseline EKG
* Hypertension that cannot be controlled by medications (>150/100 mm Hg despite optimal medical therapy).
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* Known active infection
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-07; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J George, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson, University of Texas, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- 50mg Sunitinib Malate: Sunitinib Malate 50mg capsule by mouth once daily for 4 weeks
Period: Overall Study
Arm/Group | 50mg Sunitinib Malate
Started | 30
Completed | 27
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Only study arm; treatment arm.
  Sunitinib Malate : 50mg daily x 4 weeks
Arm/Group | Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Apoptotic Indices Before and After Treatment
Description: Pathologic changes will be described using immuno-histochemical techniques (assessment of apoptotic/proliferative indices and microvessel density (MVD)) using paraffin-embedded samples and freshly cut slides from the block which are deparaffinized and rehydrated through graded alcohol, where applicable. Antigen retrieval will be accomplished by microwaving in citrate buffer from 5 to 7 minutes for the Ki-67 and MVD analysis. Mean difference in %apoptosis (measured as %TUNEL positive cells per high powered field) between pre and post treatment will be reported.
Time Frame: Baseline and 4 weeks
Population: Two patients did not complete surgery, and five patients did not have adequate tissue samples, leaving 23 patients for analysis
Measure: Mean (Standard Deviation); unit: Percentage of TUNEL positive cells
Groups:
- 50 mg Sunitinib Malate: Only study arm; treatment arm.
  Sunitinib Malate : 50mg daily x 4 weeks
Arm/Group | 50 mg Sunitinib Malate
Number analyzed (Participants) | 23
Percentage of TUNEL positive cells | -2.99 (24.42)

2. Secondary Outcome: Number of Patients Experiencing Grade ≥4 Hematologic or Grade ≥3 Non-hematologic Toxicity
Description: Adverse events were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 and were converted to version 4.0 for the purposes of ClinicalTrials.gov reporting.
Time Frame: 4 years
Measure: Number; unit: participants
Arm/Group | 50 mg Sunitinib Malate
Number analyzed (Participants) | 30
participants
  Grade >= 4 Hematologic | 1
  Grade >= 3 Non-Hematologic | 7

3. Secondary Outcome: Change in Pathologic (Microvessel Density).
Description: Pathologic changes will be described using immuno-histochemical techniques (assessment of microvessel density (MVD)) using paraffin-embedded samples and freshly cut slides from the block which are deparaffinized and rehydrated through graded alcohol, where applicable. Antigen retrieval will be accomplished by microwaving in citrate buffer from 5 to 7 minutes for the MVD analysis. Results are reported as the difference in pre and post MVD. Units for MVD are number of CD31 cells per high powered field.
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CD31 cells/High Powered Field
Arm/Group | 50 mg Sunitinib Malate
Number analyzed (Participants) | 23
CD31 cells/High Powered Field | 2.75 (7.27)

4. Secondary Outcome: Change in Systemic Parameters Before and After Sunitinib Malate Treatment.
Description: We evaluated candidate biomarkers of this pathway to predict for pharmacodynamic response to Sunitinib malate. In addition, a 7 ml plasma sample was collected at baseline and again at 4 weeks on all patients to assess possible biomarkers of response. Reported is the mean percent change in plasma concentration for each marker between 4 weeks and baseline.
Time Frame: Baseline and 4 weeks
Population: 17 patients had adequate measurements at both time points, were on an adequate dose, and took treatment at the correct time points.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 50 mg Sunitinib Malate
Number analyzed (Participants) | 17
Percent change
  ANG2 | -13.0 (28.4)
  BMP9 | -54.3 (39.6)
  CRP | 483.9 (670.0)
  D-DIMER | 14.7 (22.4)
  E-CADHERIN | -16.3 (31.3)
  E-SELECTIN | -7.9 (38.4)
  ENDOGLIN | -14.6 (16.7)
  Groa | 15.2 (44.4)
  HGF | 10.3 (33.4)
  ICAM1 | 21.9 (32.3)
  IGFBP1 | 107.6 (326.6)
  IGFBP2 | -5.9 (17.1)
  IGFBP3 | -9.8 (26.5)
  IL6 | 152.5 (277.5)
  IL8 | 90.0 (45.4)
  MCP1 | 23.6 (28.4)
  MMP2 | 0.2 (20.6)
  MMP9 | -24.2 (66.1)
  OPN | 8.8 (22.6)
  P-SELECTIN | -3.3 (96.1)
  PAI1-ACTIVE | 121.8 (157.4)
  PAI1-TOTAL | 43.2 (65.7)
  PDGF-AA | 5.8 (74.5)
  PDGF-BB | 63.8 (118.4)
  PEDF | 2.3 (26.2)
  PLGF | 500.3 (786.7)
  SDF1 | 60.6 (85.1)
  TGFB1 | -15.0 (42.2)
  TGFB2 | -10.1 (39.6)
  TGFBR3 | -8.1 (24.0)
  TSP1 | -0.9 (44.7)
  TSP2 | 9.0 (46.2)
  VCAM1 | 49.8 (68.7)
  VEGF | 135.8 (347.0)
  VEGFD | 38.6 (50.9)
  VEGFC | 2.2 (90.2)
  VEGFR1 | 14.9 (90.9)
  VEGFR2 | -30.0 (24.4)
  Tissue Factor | 190.1 (570.2)
  VWF | 60.3 (67.2)

5. Secondary Outcome: Protein Levels and Activation Status of PDGFR in Prostate Cancer Tissue.
Description: We will perform immunohistochemistry staining on snap frozen specimens for endothelial and pericyte cell staining as previously described (42). Frozen prostate tumor biopsies are sectioned at 6μm thickness and fixed with acetone for 10 minutes. Endogenous peroxidase activity is quenched with 3% hydrogen peroxide for 15 min and then blocked with 5% normal serum. The slides are incubated with the primary antibody (1;100) overnight at 4 C°, and washed with PBS. Negative controls will be included by omission of the primary antibody. Biotinylated donkey antimouse antibody (1:1000, v/v) will be applied for 30 min at room temperature, followed by application of ABC kit (Vector Lab, Inc., Burlingame, USA). Slides are again washed in PBS and the color is developed by 5 min incubation with diaminobenzidine (DAB) solution. Slides are then counterstained with hematoxylin. Mean protein levels are presented.
Time Frame: 4 years
Population: Due to changes in the field, this test was not performed due to lack of relevance.
Arm/Group | 50 mg Sunitinib Malate
Number analyzed (Participants) | 0

6. Secondary Outcome: Difference in Gene Expression Patterns Using Microarray Analysis
Description: Microarray data of 21 specimens from men enrolled who have undergone a prostatectomy and study treatment were compared to data from 21 prostatectomy only specimens. We used previously developed genomic signatures to measure the deregulation of oncogenic pathways built using Bayesian Probit models for 'metagene' factors from a singular value decomposition of top differentially expressed genes. A Monte Carlo Markov Chain was used to generate the predicted probabilities of pathway activity in normalized samples. We predicted the activity of these pathways, leading to the generation of probability measures that have previously reflected the state of pathway activity. These probability scores are interpreted as gene expression values to describe pathway activity patterns. A probability near 0 indicates a low chance of pathway activity; a probability near 1 indicates a higher likelihood of activity. Differences (treatment - control) in mean probability for each pathway are reported.
Time Frame: 4 years
Population: 21 patients had adequate samples for analysis.
Measure: Mean (Standard Deviation); unit: Probability
Arm/Group | 50 mg Sunitinib Malate
Number analyzed (Participants) | 21
Probability
  BCAT | 0.24 (0.25)
  E2F1 | 0.18 (0.25)
  PI3K | 0.14 (0.15)
  ER | 0.18 (0.33)
  MYC | 0.24 (0.23)
  IFNalpha | -0.01 (0.30)
  IFNgamma | -0.01 (0.32)
  EGFR | -0.08 (0.25)
  TGFB | -0.17 (0.30)
  STAT3 | -0.11 (0.20)
  TNFa | 0.02 (0.31)
  HER2 | 0.03 (0.24)
  RAS | 0.07 (0.16)
  HYPOXIA | 0.11 (0.25)
  AKT | -0.36 (0.19)
  SRC | -0.17 (0.16)
  P63 | -0.09 (0.17)
  Acidosis | -0.10 (0.14)
  Lactic Acidosis | -0.22 (0.20)
  P53 | 0.05 (0.17)
  PR | -0.01 (0.24)
  Glucose Deprivation | 0.11 (0.21)
  AR | 0.15 (0.20)

7. Secondary Outcome: Interstitial Fluid Pressure (IFP)
Description: Measure Interstitial fluid pressure (IFP) pre-treatment and during treatment to indirectly measure the effect of Sunitinib malate on transcapillary transport and correlate with other biologic evidence of treatment effect.Eligible patients who sign consent will undergo a baseline transrectal ultrasound (TRUS)-guided measurement of tumor IFP. Participants will then begin treatment with daily oral Sunitinib malate with biweekly monitoring for response and toxicity. After 4 weeks of therapy, patients undergo a repeat TRUS and tumor IFP measurement. Following a 1 to 2 week wash out period, patients undergo prostatectomy with pathologic tissue collection. This will be performed as a means to evaluate whether Sunitinib malate has the ability to decrease tumor IFP, and whether this correlates with other tr
Time Frame: 4 years
Population: This was an optional test and no patients chose to participate.
Arm/Group | 50 mg Sunitinib Malate
Number analyzed (Participants) | 0

8. Primary Outcome: Change in Proliferation Indices Before and After Treatment
Description: Pathologic changes will be described using immuno-histochemical techniques (assessment of apoptotic/proliferative indices and microvessel density (MVD)) using paraffin-embedded samples and freshly cut slides from the block which are deparaffinized and rehydrated through graded alcohol, where applicable. Antigen retrieval will be accomplished by microwaving in citrate buffer from 5 to 7 minutes for the Ki-67 and MVD analysis. Mean difference in %proliferation (Ki67 positive nuclei out of total nuclei) between pre and post treatment will be reported.
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Ki67 positive nuclei
Arm/Group | 50 mg Sunitinib Malate
Number analyzed (Participants) | 23
Percentage of Ki67 positive nuclei | -3.19 (6.57)

ADVERSE EVENTS:
Time Frame: 4 years
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.3.0, and have been converted to v.4.0 for entry into ClinicalTrials.gov
Arm/Group | 50 mg Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 29/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg Sunitinib Malate (N=30)
Anemia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anal mucositis (Gastrointestinal disorders) | 2
Cheilitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 13
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 11
Dysphagia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 5
Oral pain (Gastrointestinal disorders) | 5
Rectal pain (Gastrointestinal disorders) | 1
Vomitting (Gastrointestinal disorders) | 1
Chills (General disorders) | 3
Edema face (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 22
Fever (General disorders) | 3
Flu like symptoms (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Infections and infestations - Other, sinus (Infections and infestations) | 2
Infections and infestations - Other, urinary (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 13
Platelet count decreased (Investigations) | 18
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Concentration impairment (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 21
Headache (Nervous system disorders) | 6
Memory impairment (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, hair depigmentation (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other, subungual splinter hemorrhage (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other, yellowing skin (Skin and subcutaneous tissue disorders) | 10
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 4
Hypertension (Vascular disorders) | 10
Lymphedema (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes